CLINICAL TRIAL: NCT00525681
Title: The Effect of Rimonabant Treatment on Cardiovascular Risk Factors in Renal Transplant Recipients -- Pilot Safety Study
Brief Title: Interaction Between Rimonabant and Cyclosporine and Tacrolimus
Acronym: RIMONA-PILOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIMONA-PILOT
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Renal Transplantation
Keywords: Obese; Calcineurine inhibitor; Pharmacokinetics; Interaction
MeSH Terms: conditions — Obesity | interventions — Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CsA (Other): Investigation of systemic exposure of cyclosporine before and after 2 moths of co-adminiastration of rimonabant.
  Interventions: Drug: cyclosporine A
- Tac (Other): Investigation of systemic exposure of tacrolimus before and after 2 moths of co-adminiastration of rimonabant.
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: cyclosporine A — Cyclosporine is dosed twice daily and is individualized as per center practice and kept stable during the study.
  Other Names: Sandimmun Neoral
  Arms: CsA
Drug: tacrolimus — Dosing of tacrolimus is given twice daily and individualized as per center practice.
  Other Names: Prograf
  Arms: Tac

SUMMARY:
The major cause of premature death in renal transplant recipients is cardio-vascular disease. In addition, obesity is becoming a major problem in this patient population. Rimonabant does not only seem to have weight reducing properties but also weight reduction independent effects on insulin sensitivity and endothelial function, two important cardio-vascular risk factors. Rimonabant therefore is an interesting drug for the treatment of transplanted patients. Present data also indicate that rimonabant does not interact with essential immunosuppressive drugs (CsA and Tac) indicating that it most probably is safe to administer to this patient population. However this needs to be investigated in a proper manner.

DETAILED DESCRIPTION:
Renal transplant recipients are treated with life-long immunosuppressive therapy in order to prevent acute rejection episodes. The calcineurin inhibitors (CsA and Tac) are the back-bones in the immunosuppressive treatment and they have a very narrow therapeutic index. It is therefore essential to assure that new drug to be used in transplanted patients do not interact with CsA and Tac. Even though rimonabant is metabolized via the same enzyme as CsA and Tac (CYP3A4) previous in vitro and in vivo studies with relevant probe drugs in healthy volunteers do not indicate the presence of any relevant pharmacokinetic interaction. However, to be absolutely sure that it is safe to administer rimonabant in transplanted patients a 12-hour pharmacokinetic interaction investigation is included for 16 patients in the present pilot study (8 patients on CsA and 8 patients on Tac).

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipient with stable renal function (less than 20% deviation in serum creatinine the last 2 months).
* Renal transplant recipient currently on CsA or Tac and prednisolone based immunosuppression.
* BMI > 30 kg/m2 or >27 kg/m2 in combination with one or more cardio-vascular risk factors.
* > 18 years of age.
* Male patient, or female patient without childbearing potential (surgically sterilized or postmenopausal) or, if female of childbearing potential, is not lactating, has a negative pregnancy test at screening and is willing to utilize an effective method of contraception throughout the study period and for 90 Days following discontinuation of the Study Drugs.
* Signed informed consent.

Exclusion Criteria:

* Diabetes mellitus
* Severe liver disease.
* Depressive-, anxiety- or sleeping disorders.
* Estimated GFR < 25 ml/min.
* Epilepsy.
* Skin disorders that may influence laser Doppler flowmetry investigations.
* Pregnant or nursing mothers.
* Concomitant treatment with CYP3A4 inhibitors (www.cyp450.no) with interaction potential according to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Effect of rimonabant on cylosporine/tacrolimus bioavailablility | 2 months

SECONDARY OUTCOMES:
Effect of rimonabant on insulin sensitivity | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, Ph.D., Study Chair — Scholl of Pharmacy, University of Oslo
Locations (1):
- Rikshospitalet, Section of Nephrology, Oslo, Norway